CLINICAL TRIAL: NCT06209294
Title: Phase II Study on Neoadjuvant Therapy of AK104 Combined With Nab-paclitaxel/Carboplatin in Fertility Preserving Surgery for Stage IB2-IB3 Cervical Cancer (FIGO 2018)
Brief Title: Phase II Study on Neoadjuvant Therapy of AK104 Combined With Nab-paclitaxel/Carboplatin in Fertility Preserving Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xiaohua Wu (Other)
Responsible Party: Sponsor-Investigator, Xiaohua Wu, Principal Investigator, Fudan University
Organization: Fudan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NACI-CC-FSS
Record Dates: First submitted 2023-12-20; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Neoadjuvant Immunotherapy; Cervical Cancer; Fertility-sparing Surgery
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Carboplatin; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: AK104 combined with nab-paclitaxel and carboplatin (Experimental): Carboplatin, nab-paclitaxel and AK104 as neoadjuvant treatment before fertility-sparing surgery
  Interventions: Drug: AK104; Drug: Carboplatin; Drug: Nab paclitaxel

INTERVENTIONS:
Drug: AK104 — AK104(10 mg/kg) d1,22
Drug: Carboplatin — AUC=2 d1,8,15,22, 29, 36
Drug: Nab paclitaxel — 125mg／m2 d1,8,15,22,29,36

SUMMARY:
This is a Phase II study of neoadjuvant therapy of AK104 combined with nab-paclitaxel/carboplatin in fertility saving surgery for stage IB2-IB3 cervical cancer (FIGO 2018). The main questions it aims to answer are:

* · Evaluate the safety of AK104 combined with nab-paclitaxel/carboplatin in the neoadjuvant treatment of cervical cancer
* · Evaluate the tumor regression and Major Pathological Response(MPR) of AK104 combined with nab-paclitaxel/carboplatin as neoadjuvant therapy for cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign a written ICF.
* Age ≥ 18 years old and ≤ 45 years old at the time of enrollment.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Patients with histologically confirmed (2018 FIGO) stage IB2-IB3 cervical squamous cell carcinoma, adenocarcinoma, and adenosquamous carcinoma.
* Imaging evaluation showed no distant metastasis or regional lymph node metastasis, and the tumor was limited to the cervix.
* Have not received any systemic or local anti-tumor treatment for cervical cancer before the first medication, including radiotherapy, chemotherapy, immunotherapy, biological agents, small molecule targeted therapy, etc.
* Patients who require preservation of reproductive function and who are judged by the researcher to have no contraindications to childbirth surgery.
* At least 1 untreated measurable lesion according to RECIST v1.1.
* Subjects agree to collect tumor tissue and peripheral blood samples required during the screening period and research process and use them in related research.
* With good organ function:

  a) Hematology (no blood components and cell growth factor support therapy were used within 7 days before starting study treatment): i. Absolute neutrophil count ANC ≥ 1.5 × 109/L (1,500/mm3); ii. Platelet count ≥ 100 × 109/L (100,000/mm3); iii. Hemoglobin ≥ 90 g/L. b) Kidney: i. Calculated creatinine clearance* (CrCl) ≥ 50 mL/min

  * CrCl will be calculated using the Cockcroft-Gault formula (Cockcroft-Gault formula) CrCl (mL/min) = {(140 - age) × weight (kg) × 0.85}/ (serum creatinine. (mg/dL) × 72) ii .Urine protein < 2+ or 24-hour (h) urine protein quantification < 1.0 g.

  c) Liver: i. Serum total bilirubin (TBil) ≤ 1.5 × ULN ii. AST and ALT ≤ 2.5× ULN iii. Serum albumin (ALB) ≥ 28 g/L d) Coagulation function: i. International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN (e.g.

If the subject is receiving anticoagulant therapy, the subject must receive a stable dose of anticoagulant and have coagulation during screening.

Parameters (PT/INR and APTT) were within the expected range for anticoagulant therapy).

e) Heart function: i. Left ventricular ejection fraction (LVEF) ≥ 50%.

* Female subjects with childbearing potential must undergo a urine or serum pregnancy test within 3 days before taking the drug for the first time (if the urine pregnancy test result cannot be confirmed to be negative, a serum pregnancy test must be performed, and the serum pregnancy result shall prevail). and the result was negative. If a female subject of childbearing potential has sexual intercourse with a non-sterilized male partner, the subject must use an acceptable method of contraception since screening and must agree to continue using contraception methods for 120 days after the last dose of the study drug. Whether to discontinue contraception after this time point should be discussed with the investigator. Cyclic abstinence and safe period contraception are unacceptable methods of contraception.

  1. Women of childbearing potential are those who have not been surgically sterilized (i.e., bilateral fallopian tube ligation, bilateral oophorectomy, or total hysterectomy) or who have not undergone menopause (menopause is defined as at least one without alternative medical reasons). 12 consecutive months of amenorrhea and serum follicle-stimulating hormone levels within the laboratory reference range for postmenopausal women);
  2. Highly effective contraceptive methods refer to contraceptive methods that have a very low contraceptive failure rate (e.g. less than 1% per year) when used correctly and consistently. Not all birth control methods are highly effective. In addition to barrier contraceptive methods, female subjects of childbearing potential must also use hormonal contraceptive methods (such as birth control pills) alone to ensure that pregnancy does not occur.
* Subjects are willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other requirements of the study.

Exclusion Criteria:

* The histopathological types are small cell carcinoma, gastric adenocarcinoma, etc.
* In addition to cervical cancer, subjects suffered from other malignant tumors within 3 years before enrollment. Subjects with other malignant tumors that have been cured by local treatment, such as basal or cutaneous squamous cell carcinoma, superficial bladder cancer, breast cancer, etc., are not excluded.
* Enroll in another clinical study at the same time, unless it is an observational, non-interventional clinical study or the follow-up period of an interventional study.
* Patients with distant tumor metastasis or local and regional lymph node metastasis.
* Patients who received non-specific immunomodulatory therapy (such as interleukins, interferons, thymosin, tumor necrosis factor, etc., excluding IL-11 used to treat thrombocytopenia) within 2 weeks before the first medication; Received non-specific immunomodulatory therapy within 1 week before the first medication Chinese herbal medicine or Chinese patent medicine with anti-tumor indications.
* Suffering from active autoimmune diseases that require systemic treatment (such as disease-modifying drugs, corticosteroids, immunosuppressive treatment), Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a systemic therapy.
* Patients have a history of non-infectious pneumonia or pneumonia requiring systemic glucocorticoid treatment or a current history of interstitial lung disease.
* With a history of severe bleeding tendency or coagulation disorder.
* Patients with currently uncontrolled comorbid diseases, including but not limited to decompensated cirrhosis, nephrotic syndrome, uncontrolled metabolic disorders, severe active peptic ulcer disease or gastritis, or a mental illness/social condition that would limit the subject's ability to comply with research requirements or affect the subject's ability to provide written informed consent.
* Patients with history of myocarditis, cardiomyopathy, and malignant arrhythmia. Patients suffered unstable angina, congestive heart failure or vascular disease requiring hospitalization (such as aortic aneurysm or peripheral venous thrombosis requiring surgical repair) within 12 months before the first dose, or other heart damages (such as poorly controlled arrhythmia, myocardial infarction or ischemia) that may affect the safety evaluation of the study.

Patients with a history of esophageal and gastric varices, severe ulcers, unhealed wounds, gastrointestinal perforation, abdominal fistula, gastrointestinal obstruction, intra-abdominal abscess or acute gastrointestinal bleeding within 6 months before the first administration; Patients suffered any arterial thromboembolic event, NCI CTCAE version 5.0 grade 3 or above, venous thromboembolism, transient ischemic attack, cerebrovascular accident, hypertensive crisis or hypertensive encephalopathy within 6 months before the first dose; Patients with acute exacerbation of COPD within 1 month before first dose; Current hypertension with systolic blood pressure ≥160mmHg or diastolic blood pressure ≥100mmHg after treatment with oral antihypertensive drugs.

* Patients with active or clear history of inflammatory bowel disease (such as Crohn's disease, ulcerative colitis or chronic diarrhea).
* Patients with serious infection occurring within 4 weeks before the first dose, including but not limited to complications requiring hospitalization, sepsis or severe pneumonia; Patients with active infection (excluding antiviral therapy for hepatitis B or hepatitis C) that has been treated with systemic anti-infectious therapy within 10 days before the first dose.
* Patients suffered major surgery or serious trauma within 30 days before the first medication; or minor local surgery within 3 days before the first medication (excluding central venous catheterization via peripheral venipuncture).
* Patients with a history of immunodeficiency; those with positive HIV antibody test; Patients who are taking long-term systemic corticosteroids or other immunosuppressants.
* Subjects who are known to have active pulmonary tuberculosis (TB) and are suspected of having active TB need to undergo clinical examination to exclude (such as sputum tuberculosis bacilli examination, chest X-ray, etc.); known active syphilis infection.
* Patients with history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
* Subjects with untreated active hepatitis B (HBsAg positive and HBV-DNA exceeding 1000 copies/ml (200 IU/ml) or higher than the lower limit of detection).Subjects with hepatitis B are required to receive anti-hepatitis B virus treatment during the study treatment period; subjects with active hepatitis C (HCV antibody positive and HCV-RNA levels above the lower limit of detection).
* Patients who have received a live vaccine within 30 days before the first dose, or plan to receive a live vaccine during the study.
* Patients who are hypersensitive to any component of any study drug; with history of severe hypersensitivity reactions to other monoclonal antibodies.
* Patients with history of mental illness, substance abuse, alcoholism, or drug abuse.
* Pregnant or lactating women.
* Patients with any past or current disease, treatment, or laboratory test abnormality may confuse the research results and affect the subject's full participation in the research, or participation in the research may not be in the best interests of the subject.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Up to approximately 6 mouths
  To evaluate the safety of AK104 combined with nab-paclitaxel and carboplatin in the neoadjuvant treatment of cervical cancer
Tumor regression rate | within 14 working days after operation
  The change of tumor size after the treatment,
Objective response rate | 4-6 weeks after the second cycle(21 days per cycle) of neoadjuvant treatment
  Objective response rate is the proportion of subjects with complete response(CR) or partial response(PR) , based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
The success rate of fertility sparing surgery | Up to approximately 6 mouths
  The rates of patients who can successfully preserve fertility.

SECONDARY OUTCOMES:
Major pathological response (MPR) rate | within 14 working days after operation
  MPR rate is defined as the percentage of participants having ≤ 10% viable tumor cells in the pathological examination of resected specimens.
Pathological Complete Response (pCR) rate | within 14 working days after operation
  pCR rate is defined as the percentage of participants lacking of evidence of viable tumor cells in the pathological examination of resected specimens.
Progression-free survival | Nearly 5 years after treatment
  Survival of patients
Overall survival | Nearly 5 years after treatment
  Overall survival of patients
Pregnant rates | Nearly 5 years after treatment
  Pregnant rates of patients after treatment

OTHER OUTCOMES:
Ratio of different immune cells in tumor micro-environment after neoadjuvant treatment | Up to approximately 6 mouths
  Biomarkers associated with efficacy of neoadjuvant immune-chemotherapy after the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Data is available per require after approved by ethics broad